CLINICAL TRIAL: NCT06079580
Title: Examination of Multifidus Muscle and Balance in Lumbar Spinal Stenosis
Brief Title: Patients With Lumbar Spinal Stenosis With Balance Disorder
Status: Completed | Type: Observational
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Musa Güneş, Study director, PT, MsC, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Karabuk University
Other Study IDs: Karabuk University-01
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Lumbar spinal stenosis with balance disorders: According to the single-leg balance test, patients who maintain static balance for less than 10 seconds will be grouped as having impaired balance.
- Patients with Lumbar spinal stenosis with normal balance: According to the single-leg balance test, patients who maintain their static balance for more than 10 seconds will be grouped as having normal balance.

SUMMARY:
It is seen that patients with Lumbar Spinal Stenosis often experience balance problems. Although the relationship between muscle thickness and balance has been explained, there are insufficient studies investigating the relationship between balance problems and muscle thickness in patients with LSS. In addition, no study has been found comparing the difference in muscle thickness and cross-sectional area in LSS patients with poor and normal balance. In addition, in LSS, pain, disability and fear of falling in balance disorders are nor clear. The aim of our study is to examine the relationship between balance and biopsychosocial factors that can affect it.

DETAILED DESCRIPTION:
The stability and balance of the lumbar spine depends on the paraspinal muscles surrounding it. In addition, the atrophy of the muscle in this area leads to deterioration of the body's stability. The multifidus muscle is important for the lumbar region due to its multiple connections. Today, morphological factors of paraspinal muscles are being investigated. The degeneration occurring in these muscles also causes a decrease in the thickness and cross-sectional areas of the muscle. This condition is associated with loss of balance in various populations. However, this relationship has not been adequately investigated in patients with lumbar spinal stenosis. At the same time, the intensity of pain affects balance and causes disruptions. Balance problems in older adults can lead to falls, leading to vertebral and femoral neck fractures. These injuries cause a decrease in quality of life. When the literature is examined, it is seen that patients with LSS often have balance problems. Parameters such as muscle mass, pain, disability and fear of falling affect this factor. However, although the relationship between muscle thickness and balance has been described in various populations, there are insufficient studies investigating the relationship between balance problems and muscle thickness in patients with LSS. In addition, no study has been found comparing the difference in muscle thickness and cross-sectional area in LSS patients with poor and normal balance. In addition, it is observed that biopsychosocial factors such as pain, disability and fear of falling in balance disorders are not adequately explained. In this context, our study aims to The aim of our study is to examine the relationship between balance and biopsychosocial factors that can affect it.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with L4/5 lumbar spinal stenosis by MRI,
* Patients who can stand independently
* Volunteering to participate in the study

Exclusion Criteria:

* Patients who did not agree to participate in the study,
* Having a history of serious neurological diseases such as Parkinson's, hemiplegia, multiple sclerosis,
* Having undergone a surgical operation on the lumbar region within the last year,
* Having severe joint disorders in the lower extremities,
* Having malignancy in the spine,
* Having had an operation on the lower extremity,
* Having vision and/or vestibular system problems,
* Those who do not cooperate well

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Lumbar Spinal Stenosis
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Static balance | First Day
  The static balance of the patients will be evaluated with the 'Single Leg Standing Balance Test'.

SECONDARY OUTCOMES:
Dynamic balance | First day
  The dynamic balance of the patients will be evaluated with the 'Timed Up and Go Test (TUG)'.
Pain Severity | First day
  Evaluation of individuals' back and leg pain intensity will be done with the 'Numeric Rating Scale'.
Disability | First day
  Oswestry Disability Index will be used to evaluate the degree of loss of function that occurs with low back pain.
Faling | First day
  Fear of falling will be assessed with the International Fall Efficacy Scale (FES-I).
Muscle thickness | First day
  Multifidus muscle thickness at the L4/5 level will be evaluated using an MRI device.
Muscle cross-sectional area | First day
  Multifidus muscle cross-sectional area at the L4/5 level will be evaluated using an MRI device.

CONTACTS AND LOCATIONS:
Locations (1):
- Karabuk University, Physiotherapy and Rehabilitation Application and Research Center, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farrokhi MR, Haghnegahdar A, Rezaee H, Sharifi Rad MR. Spinal sagittal balance and spinopelvic parameters in patients with degenerative lumbar spinal stenosis; a comparative study. Clin Neurol Neurosurg. 2016 Dec;151:136-141. doi: 10.1016/j.clineuro.2016.10.020. Epub 2016 Oct 31. PMID 27842292
- [Background] Thornes E, Robinson HS, Vollestad NK. Dynamic balance in patients with degenerative lumbar spinal stenosis; a cross-sectional study. BMC Musculoskelet Disord. 2018 Jun 15;19(1):192. doi: 10.1186/s12891-018-2111-x. PMID 29902972
- [Background] Ito T, Sakai Y, Yamazaki K, Oikawa M, Morita Y. Relationship Between L4/5 Lumbar Multifidus Cross-Sectional Area Ratio and Fall Risk in Older Adults with Lumbar Spinal Stenosis: A Retrospective Study. Geriatrics (Basel). 2019 Jun 21;4(2):38. doi: 10.3390/geriatrics4020038. PMID 31234297